CLINICAL TRIAL: NCT04133571
Title: Bladder Irrigation With 0.05% Lidocaine Normal Saline Solution for Prevent Postoperative Catheter Related Bladder Discomfort (CRBD) Under ANI Monition After Transurethal Surgery
Brief Title: Bladder Irrigation 0.05% Lidocaine Decreases Postoperative CRBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chia-Heng Lin, MD, Physician, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-F(I)-20190065
Record Dates: First submitted 2019-09-01; First posted 2019-10-21 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Bladder Discomfort
Keywords: catheter-related bladder discomfort; lidocaine
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Control group: using normal saline for bladder irrigation
- Study group (Experimental): Study group: using 0.05% Lidocaine normal saline solution for bladder irrigation
  Interventions: Drug: 0.05% Lidocaine

INTERVENTIONS:
Drug: 0.05% Lidocaine — 0.05% lidocaine with normal saline as a bladder irrigation solution after transurethral surgery intravenous pethidine to decrease CRBD if needed
  Other Names: intravenous pethidine 0.25 mg/kg
  Arms: Study group

SUMMARY:
Catheter-related bladder discomfort (CRBD) secondary to an indwelling urinary catheter is very distressing, and it may get worse in patients undergoing transurethral surgery for damage urethra by a surgical instrument as well as a sizable and urinary catheter placement. Lidocaine, a local anesthetic, showed of analgesic, sedative, and anti-inflammatory effect. Therefore, the investigators prepared a 0.05% lidocaine in normal saline as a bladder irrigation solution after surgery to reduce Catheter-related bladder discomfort.

DETAILED DESCRIPTION:
Catheter-related bladder discomfort (CRBD) secondary to an indwelling urinary catheter is very distressing. It is not unusual that patients who have been catheterized under anesthesia complain of an urge to void in the postoperative period because of catheter-related bladder irritation. Bladder catheterization induces bladder irritation whose symptoms (urge to void and discomfort in the suprapubic region) are similar to the symptoms of an overactive bladder (urinary frequency and urgency with or without urge incontinence), caused by involuntary contractions of the bladder mediated by muscarinic receptors. The discomforts are quickly getting worse in patients undergoing transurethral surgery by a surgical instrument as well as a sizable urinary catheter placement. Recently, antimuscarinic drugs for treat overactive bladder, such as tolterodine and oxybutynin, have been tried for prevention of CRBD with variable success. However, they may cause side effect including palpitation, dry mouth, drowsiness, dizziness or headache. Lidocaine, a local anesthetic, showed of analgesic, sedative and anti-inflammatory effect. Therefore, the investigators prepared a 0.05% lidocaine in normal saline as a bladder irrigation solution after surgery to reduce Catheter-related bladder discomfort.

Objectives:

The aim of this study were:

1. to evaluate the efficacy to prevent CRBD with Bladder irrigation with 0.05% Lidocaine normal saline solution
2. to observe the change of vital sign with Bladder irrigation with 0.05% Lidocaine normal saline solution
3. to see the side effect of with Bladder irrigation with 0.05% Lidocaine normal saline solution

ELIGIBILITY:
Inclusion Criteria:

* Patients who received regular transurethral surgery were inserted left foley catheter for urine drainage or bladder irrigation.
* American Society of Anesthesiologists(ASA)class:Ι-Ⅲ
* Age:20-70years
* Sex:Male

Exclusion Criteria:

* Lidocaine allergy
* cardiac conduction with partial or total block
* patient with progressive hepatic or renal impairment
* patient with class III anti-arrhythmia agent(ex:amiodarone)
* patient with acute porphyria

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-05-17 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
using Numerical rating scale to measure pain alleviate | 6 hours
  measurement of numerical pain rating scale from 0 (no pain): no pain to 10 (severe pain intolerable) as maintain the score of analgesia nociception index within 50-70 ( over 70 may need to evaluate analgesia overdose and under 50 to evaluate pain or hemodynamic changes)
using catheter-related bladder discomfort score to evaluate CRBD alleviation | 6 hours
  measurement of catheter-related bladder discomfort score (grade 1: none, grade II: mild, grade III: moderate, grade IV: severe

SECONDARY OUTCOMES:
using the sphygmomanometer to monitor blood pressure | 6 hours
  monitoring fluctuate systolic, diastolic blood pressure(unit: mmHg)
checking the heart rate of patient by the pulse oximeter | 6 hours
  checking the heart rate(unit: the heart beats per minute) by the pulse oximeter
monitoring the hemodynamic changes by using the analgesia nociception index(ANI) | 6 hours
  maintain the score of analgesia nociception index within 50-70 ( over 70 may need to evaluate analgesia overdose and under 50 to evaluate pain or hemodynamic changes) and observe the changes under the situation of discomfort and pain
checking the physiological response, vomiting or not | 6 hours
  checking vomiting or not
measure the physiological response to the hypothermia of patient | 6 hours
  measure if the temperature below 35.0°C so called the hypothermia(unit: °C) of patient by the thermometer
measuring the amount of oxygen in the blood | 6 hours
  check SaO2(arterial oxygen saturation) by the pulse oximeter(unit: %), a small beams of light pass through the blood in the finger, measuring the amount of oxygen, should maintain in 90%-100%
assess the electrolyte imbalance by checking the content of Na | 6 hours
  assess the electrolyte imbalance, maintain Na(unit: mmol/L) in 135-145, by 2 to 5 ml of blood testing
assess the electrolyte imbalance by checking the content of K | 6 hours
  assess the electrolyte imbalance, maintain K(unit: mmol/L) in 3.5-5.1, by 2 to 5 ml of blood testing
assess the electrolyte imbalance by checking the content of Ca++ | 6 hours
  assess the electrolyte imbalance, maintain Ca++(unit: mg/dL) in 4.6~5.32, by 2 to 5 ml of blood testing

CONTACTS AND LOCATIONS:
Overall Officials: Chia-heng Lin, MD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan